CLINICAL TRIAL: NCT06608043
Title: Reborn Lifestyle Adjustment Program for Breast Cancer Patients
Brief Title: Reborn Lifestyle Adjustment Program
Status: Recruiting | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Other Study IDs: E-22686390-050.99-46613
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Occupational Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention Group: This intervention group consists of multi-component modules developed to help individuals with breast cancer adopt a healthy lifestyle and improve their quality of life. The sessions are based on the 'Do Live Well' model, Kolb's Experiential Learning Theory, and CBT-based problem-solving skills.
  Interventions: Behavioral: Reborn lifestyle adjustment program
- Control Group: Patients in the control group will continue conventional medical treatments, occupational therapy and physiotherapy sessions.
  Interventions: Procedure: Conventional Physiotherapy and Occupational Therapy

INTERVENTIONS:
Behavioral: Reborn lifestyle adjustment program — The sessions are based on the 'Do Live Well' model, Kolb's Experiential Learning Theory, and CBT-based problem-solving skills.
  Introduction to the Reborn Lifestyle: Core principles of the Reborn Program for building a healthy lifestyle during and after breast cancer.
  Physical Activity: The role of physical activity during treatment and exercises to boost energy levels.
  Fatigue Management: Scientific methods for managing fatigue during and after treatment.
  Pain Management: Effective techniques to reduce pain and improve quality of life.
  Mental Health Burden: Strategies to alleviate mental health burdens and cope with stress.
  Quality Sleep: Practical methods to improve sleep patterns and achieve quality rest.
  Preventive Rehabilitation Approaches: Essential rehabilitation strategies to protect health and reduce recurrence risk.
  The study will be conducted online, with evaluations and sessions via Zoom before and after the 12-week modules.
  Groups: Intervention Group
Procedure: Conventional Physiotherapy and Occupational Therapy — Patients in the control group will continue conventional medical treatments, occupational therapy and physiotherapy sessions.
  Groups: Control Group

SUMMARY:
The aim of this study is to investigate the effects of the reborn lifestyle regulation program on physical activity, fatigue level, pain, mental health burden and quality of life in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Being a female individual aged 18 or older
* Have been diagnosed with Stage I, II, or III breast cancer
* At least 6 months have passed since the completion of chemotherapy
* Approval by an oncologist to participate in the study
* Having internet access and the ability to connect online
* Scoring above 23 on a standardized Mini Mental Status Examination Test
* Being in the contemplation stage according to the Transtheoretical Model

Exclusion Criteria:

* Having a neurological or systemic disease that could significantly affect the course of the intervention
* Having metastasis that could impact the sustainability of the study
* Suffering from neuropathic pain
* Having participated in a healthy lifestyle program within the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer Specific Quality of Life Scale | 12 weeks
  An adjunct to the EORTC QLQ-C30, this scale assesses breast cancer-specific symptoms and treatment-related side effects. It includes subscales for body image, sexual function, and treatment side effects, rated on a 4-point Likert scale. The Turkish version was adapted by Demirci et al. in 2011.
Modified Borg Scale | 12 weeks
  Developed by Borg in 1970, this unidirectional scale (0-10) measures the effort exerted during physical exercise, particularly in assessing dyspnea severity. Participants rate their dyspnea over the past week, with "0" indicating no shortness of breath and "10" indicating severe shortness of breath.
Sit up Test | 12 weeks
  This test measures leg strength and endurance by counting how many times a participant can sit and stand from a chair within 30 seconds. A score of fewer than 10 sit-ups indicates lower extremity weakness. The Turkish validity and reliability were established by Demir and Öztürk in 2020.
Cancer Fatigue Scale | 12 weeks
  The CFS, developed by Okuyama et al. (2000) and validated in Turkish by Şahin et al. (2018), evaluates fatigue in individuals with cancer across three domains: physical, emotional, and cognitive. The scale consists of 15 items, rated on a Likert scale from 1 (not at all) to 5 (very much).
McGill-Melzack Pain Questionnaire | 12 weeks
  Developed by Melzack in the 1970s and validated in Turkish by Kuguoglu et al. (2003), the MPQ assesses the quality and intensity of pain through four sections, including sensory and perceptual dimensions. Scores range from 0 to 112, with higher scores indicating more severe pain.
Depression Anxiety Stress Scale (DASS-21) | 12 weeks
  The DASS-21, developed by Lovibond & Lovibond (1995) and validated in Turkish by Sarıçam (2018), assesses mental health across three dimensions: depression, anxiety, and stress. Each dimension consists of 7 items rated on a 4-point Likert scale. Higher scores indicate more severe symptoms.
Pittsburgh Sleep Quality Index (PSQI) | 12 weeks
  Developed by Buyyse et al. (1989) and validated in Turkish by Agargun et al., the PSQI assesses sleep quality over the past month across seven components. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Scale | 12 weeks
  This 30-item scale assesses the quality of life in cancer patients across three domains: global health, functional, and symptoms. Higher scores in functional and general health indicate better well-being, while higher symptom scores indicate more severe issues.
University of Rhode Island Scale for Assessing Change | Baseline
  This scale assesses individuals' readiness for change as part of the study's inclusion criteria. Developed by Prochaska et al. (1983), it consists of 32 items rated on a 5-point Likert scale. The scale has 4 sub-dimensions: pre-contemplation, contemplation, action, and maintenance. The Turkish validity and reliability were confirmed by Menekli and Fadiloglu (2012). Higher scores indicate a more positive attitude toward change.
Mini Mental Status Examination Test | Baseline
  The MMSE will be used to determine cognitive levels for study inclusion. Developed by Folstein et al. in 1975, this tool assesses cognitive performance across five domains. The test is widely used due to its ease and quick administration. Scores range from 0 to 30, with a cut-off of 23/24, as validated in Turkish by Gungen et al.
Visual Analog Scale | 12 weeks
  The VAS, developed by Hayes and Patterson (1921) and validated in Turkish by Aydın et al. (2011), is used to measure pain severity. A 10 cm line is marked from "no pain" to "unbearable pain," and the patient places a mark according to their pain level.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Ondes, MSc, Study Chair — Atlas University
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No